CLINICAL TRIAL: NCT07018622
Title: Effect of Sodium-Glucose Cotransporter 2 Inhibition on Urinary Biomarkers of Kidney Injury After Platinum-Based Chemotherapy
Brief Title: Protecting the Kidney's Proximal Tubules From Platinum-Based Chemotherapy Toxicity
Acronym: DAPA-ARMOR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NMM-5274
Record Dates: First submitted 2025-05-26; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors; Cisplatin Nephrotoxicity
Keywords: Solid Tumors; Platinum-Based Chemotherapy; Cisplatin; Carboplatin; Nephrotoxicity; Kidney Tubules, Proximal; SGLT2 Inhibitors; Kidney Injury Molecule-1; Renal Protection; Chemotherapy-Induced Kidney Injury; Randomized Controlled Trial; Urinary Biomarkers; Dapagliflozin
MeSH Terms: interventions — dapagliflozin; olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): This arm aims to evaluate the potential nephroprotective effect of SGLT2 inhibition using urinary biomarkers of tubular injury.
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet
- Placebo (Placebo Comparator): This group serves as a control to evaluate the efficacy and safety of dapagliflozin in preventing platinum-induced nephrotoxicity.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 MG Oral Tablet — Participants in this arm will receive oral dapagliflozin 10 mg daily starting one day before platinum-based chemotherapy infusion (cisplatin or carboplatin) and continuing for 72 hours. The intervention aims to assess the potential nephroprotective effect of SGLT2 inhibition. Standard supportive care including hydration and magnesium supplementation will be provided to all participants.
  Other Names: Forxiga; AZD2281
  Arms: Dapagliflozin
Drug: Placebo Oral Tablet — Participants in this arm will receive a matched oral placebo starting one day before platinum-based chemotherapy infusion (cisplatin or carboplatin) and continuing for 72 hours. Standard supportive care including hydration and magnesium supplementation will also be provided. Investigators and participants will remain blinded to the group assignments.
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
Patients with cancer who receive platinum-based chemotherapy are at increased risk of kidney injury caused by these drugs. This form of toxicity can lead to treatment delays, dose reductions, or permanent discontinuation of chemotherapy, all of which can negatively impact cancer outcomes and increase patient morbidity. Despite the clinical significance, there are currently no effective strategies to prevent platinum-induced kidney damage. Existing preventive measures-such as hydration, mannitol use, and magnesium supplementation-are limited and not always effective.

This clinical trial investigates whether a type of medication known as a Sodium-Glucose Cotransporter 2 (SGLT2) inhibitor, specifically dapagliflozin, can protect the kidneys from damage during platinum-based chemotherapy in patients with solid tumors. Researchers believe that blocking SGLT2 in the kidney may reduce toxicity in the proximal tubules-the area most affected by platinum drugs.

The primary goal of this study is to compare the levels of a specific urinary biomarker of kidney injury (called KIM-1) 72 hours after chemotherapy, between patients who receive dapagliflozin and those who receive a placebo. Lower levels of this biomarker may indicate that dapagliflozin is helping protect the kidneys.

Secondary goals include comparing additional urinary biomarkers of kidney damage and function-such as EGF (epidermal growth factor), N-acetyl-β-D-glucosaminidase (uNAG), albumin (AlbU), and β2-microglobulin (uβ2-m)-at 72 hours and 7 days after chemotherapy. The study will also assess:

The percentage of patients who develop acute kidney injury, Changes in estimated glomerular filtration rate (a measure of kidney function), Electrolyte abnormalities (sodium, magnesium, phosphorus), And any adverse events associated with dapagliflozin use. As exploratory objectives, the trial will also evaluate cancer treatment response between groups (using RECIST 1.1 criteria) and the overall safety and tolerability of dapagliflozin compared to placebo.

This is a randomized, double-blind, placebo-controlled clinical trial, meaning that participants will be randomly assigned to receive either dapagliflozin or a placebo, and neither the patients nor the study team will know who receives which treatment until the study ends.

The central hypothesis is that dapagliflozin will reduce urinary biomarkers of kidney injury by at least 50% compared to placebo, offering a potential protective strategy against platinum-induced nephrotoxicity without interfering with cancer treatment.

DETAILED DESCRIPTION:
Platinum-based chemotherapy agents such as cisplatin and carboplatin are widely used in the treatment of various solid tumors due to their efficacy. However, their clinical utility is frequently limited by nephrotoxicity, predominantly targeting the proximal tubular epithelium. This can lead to acute kidney injury (AKI), electrolyte imbalances (notably hypomagnesemia, hyponatremia, and hypophosphatemia), and progression to chronic kidney disease (CKD). Current preventive strategies are largely supportive and include aggressive hydration, mannitol-induced diuresis, and magnesium supplementation, none of which offer specific cellular protection.

Recent evidence suggests that inhibitors of the sodium-glucose cotransporter type 2 (SGLT2 inhibitors or iSGLT2s), such as dapagliflozin, may confer renal protective effects beyond their original indication for type 2 diabetes mellitus. Mechanistically, SGLT2 inhibition reduces proximal tubular reabsorption of sodium and glucose, leading to improved tubular oxygenation and reduced inflammatory and oxidative stress signaling. This has been associated with reduced progression of CKD and favorable modulation of tubular injury markers in both diabetic and non-diabetic populations.

The present study, DAPA-ARMOR, is a randomized, double-blind, placebo-controlled clinical trial designed to assess the nephroprotective effects of dapagliflozin in adult patients with solid tumors undergoing platinum-based chemotherapy. The hypothesis is that short-term prophylactic administration of dapagliflozin can reduce proximal tubular injury, as evidenced by changes in urinary biomarkers.

The primary endpoint is the difference in urinary levels of Kidney Injury Molecule-1 (KIM-1) 72 hours after platinum administration, between the intervention (dapagliflozin) and control (placebo) arms.

Secondary endpoints include changes in additional urinary biomarkers associated with tubular injury and repair:

uEGF (urinary Epidermal Growth Factor) uNAG (N-acetyl-β-D-glucosaminidase) uAlb (urinary albumin) uβ2-microglobulin These biomarkers will be measured at baseline, 72 hours (±3 days), and 168 hours (±7 days) after chemotherapy administration.

Additional secondary endpoints include:

Incidence of AKI at 72 hours and 7 days post-chemotherapy (defined per KDIGO criteria), Changes in estimated glomerular filtration rate (eGFR) using the CKD-EPI 2021 equation (Cystatin C and creatinine-based), Incidence of chemotherapy-related electrolyte disturbances (Na, Mg, P), Frequency and severity of adverse events graded according to the CTCAE (Common Terminology Criteria for Adverse Events).

Exploratory outcomes will assess:

Cancer response rate using RECIST 1.1 criteria at the first post-randomization imaging evaluation, Tolerability of dapagliflozin during chemotherapy. The study drug (dapagliflozin) or placebo will be administered starting 24 hours prior to platinum chemotherapy and continued for a total of 4 days, covering the period of expected peak tubular exposure and injury.

Participants will be stratified by type of platinum agent used. Urine and blood samples will be collected at pre-specified timepoints for biomarker analysis and laboratory monitoring.

The study design aims to ensure high internal validity while capturing clinically relevant endpoints that could inform future strategies to mitigate chemotherapy-induced nephrotoxicity without compromising oncologic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Diagnosis of a solid tumor requiring a platinum-based chemotherapy regimen (cisplatin or carboplatin)
* Expected survival > 4 months
* ECOG performance status 0-2

Exclusion Criteria:

* History of nephrectomy
* History of kidney transplant
* Concurrent use of known nephrotoxic drugs (e.g., aminoglycosides, amphotericin B, cyclophosphamide, ifosfamide, methotrexate)
* Type 1 diabetes mellitus
* Poorly controlled type 2 diabetes (HbA1c > 8% or fasting glucose > 200 mg/dL in the past month)
* Active glomerulopathy
* Prior use of SGLT2 inhibitors or current indication for their use
* eGFR < 20 ml/min/1.73 m²
* Active urinary tract infection
* Unresolved obstructive uropathy
* Participation in another clinical trial
* History of recurrent genitourinary infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Urinary KIM-1/Creatinine (uKIM-1/Cr) expression at 72 hours | 72 hours (Day 3) after platinum administration
  Measurement of urinary KIM-1 normalized to creatinine (uKIM-1/Cr [pg/mg]) to evaluate renal tubular injury at 72 hours after platinum-based chemotherapy, comparing dapagliflozin vs. placebo.

SECONDARY OUTCOMES:
Urinary Epidermal Growth Factor levels adjusted by creatinine (EGF/Cr) | Baseline to Day 3 and Day 7
  Quantification of urinary EGF concentration adjusted by urinary creatinine (uEGF/Cr [ng/mg Cr]) as a marker of tubular function at 0, 72 hours (Day 3) and 168 hours (Day 7) following platinum-based chemotherapy. The analysis will compare mean absolute values and changes from baseline between the dapagliflozin and placebo groups.
Urinary N-acetyl-β-D-glucosaminidase levels adjusted by creatinine (uNAG/Cr) | Baseline to Day 3 and Day 7
  Measurement of urinary uNAG activity adjusted by urinary creatinine (uNAG/Cr [U/g]) to assess proximal tubular injury at 72 hours (Day 3) and 168 hours (Day 7) following platinum-based chemotherapy. The analysis will compare mean absolute values and changes from baseline between the dapagliflozin and placebo groups.
Urinary Albumin levels adjusted by creatinine (AlbU/Cr) | Baseline to Day 3 and Day 7
  Determination of urinary albumin excretion adjusted by urinary creatinine (AlbU/Cr [mg/g]) as an indicator of glomerular and tubular dysfunction at 72 hours (Day 3) and 168 hours (Day 7) post-chemotherapy. The analysis will compare mean absolute values and changes from baseline between the dapagliflozin and placebo groups.
Urinary β2-microglobulin levels adjusted by creatinine (uβ2-m/Cr) | Baseline to Day 3 and Day 7
  Assessment of urinary β2-microglobulin concentration adjusted by urinary creatinine (uβ2-m/Cr [mg/g]) to evaluate proximal tubular injury at 72 hours (Day 3) and 168 hours (Day 7) following platinum-based chemotherapy. The analysis will compare mean absolute values and changes from baseline between the dapagliflozin and placebo groups.
Urinary Kidney Injury Molecule-1 levels adjusted by creatinine (KIM-1/Cr) | Baseline to day 7 after platinum administration
  Quantification of urinary KIM-1 concentration adjusted by urinary creatinine (uKIM-1/Cr [pg/mg]) as a biomarker of renal tubular injury at baseline (pre-chemotherapy), and 168 hours (Day 7) following platinum-based chemotherapy. The analysis will compare mean absolute values and changes from baseline between the dapagliflozin and placebo groups.
Incidence of Acute Kidney Injury (AKI) at 72 hours and Day 7 | Baseline to Day 3 and Day 7
  Comparison of the proportion of participants developing acute kidney injury (AKI) [KDIGO criteria] at 72 hours and 7 days post-platinum chemotherapy with and without dapagliflozin.
Estimated Glomerular Filtration Rate (eGFR) at 72 hours and Day 7 | 72 hours (Day 3), 168 hours (Day 7) after platinum administration
  Comparison of the estimated glomerular filtration rate (eGFR) (using CysC-Cr CKD-EPI 2021 formula) at 72 hours and 7 days after platinum chemotherapy, with and without dapagliflozin.
Safety and tolerability of dapagliflozin in patients with solid tumors receiving platinum-based chemotherapy | From first dose of study drug through 4 weeks of follow-up
  Monitoring and comparison of adverse events as graded by CTCAE v5.0, with a focus on severity including withdrawal or dose interruption, comparing dapagliflozin vs. placebo.

OTHER OUTCOMES:
Electrolyte abnormalities (sodium, magnesium, phosphorus) at 72 hours and Day 7 | 72 hours (Day 3), 168 hours (Day 7) after platinum administration
  Comparison of the proportion of patients with alterations in sodium, magnesium, and/or phosphorus levels at 72 hours and 7 days after platinum chemotherapy, with and without dapagliflozin.
Oncologic response by RECIST 1.1 criteria | Up to 24 weeks post-randomization
  Comparison of tumor response between groups using RECIST 1.1 criteria from randomization to the first oncologist-requested imaging evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Mejía-Vilet, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", México, Tlalpan, Mexico